CLINICAL TRIAL: NCT05255848
Title: Role of Nebulized Heparin in Non-severe and Severe Covid-19 Patients Admitted to COVID Complex LRH, MTI: A Randomized Controlled Trial
Brief Title: Nebulised Heparin in Patients With COVID-19 Pneumonia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lady Reading Hospital, Pakistan (Other Government)
Responsible Party: Principal Investigator, Muhammad Imran, Registrar Pulmonology Unit (Principal Investigator), Lady Reading Hospital, Pakistan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 294/LRH/MTI
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Nebulised Heparin; ARDS; Intubation; Mortality
MeSH Terms: conditions — COVID-19 | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Heparin sodium will be administered as a nebulised aerosol dose of 5000 IU heparin three times a day (TDS) via an ai compressor nebuliser plus standard of care treatment
  Interventions: Drug: Unfractionated heparin
- No Intervention (No Intervention): Participants assigned to 'standard care' will receive the standard care required as determined by the treating team and will not be treated with nebulised heparin

INTERVENTIONS:
Drug: Unfractionated heparin — Patients will be given the same standard of care treatment plus nebulized heparin 5000IU every 8 hours started 24 hours after randomization, using a compressed air nebulizer, and will be continued for one week. In case of any complication, if the attending physician feels it necessary intervention treatment will be stopped
  Arms: Intervention

SUMMARY:
While the pandemic continues to incite panic and the guideline recommendations regarding management of COVID continue to change, we have growing evidence that ARDS secondary to Covid-19 is associated with disseminated intravascular and alveolar fibrin deposition1. Strategies devised to reduce mucous and fibrin plugs will greatly help in preventing patients from progressing to invasive ventilation2 which if happens will obviously overburden the compromised intensive care facilities. Offering heparin in nebulized form has greatly reduced levels of coagulation activation in the lungs both in animal studies and in patients with acute lung injury3. As Heparin prevents further fibrin deposition but is ineffective in the removal of pre-existing fibrin plug, so early use of heparin during the course of the disease may help in limiting the complications of ARDS and hence reducing the burden faced by our intensive care units.

A prospective randomized controlled trial will be carried out in patients admitted to COVID complex to see its effects on disease progression and its role in preventing patients from progressing to require Invasive Mechanical Ventilation while being administered through local route rather than systemic. Moreover, it will also give insight and way forward regarding the improvement in the survival and earlier discharge

DETAILED DESCRIPTION:
Second-year into the deadly COVID-19 pandemic and humanity continues to get affected/infected. The world has seen a total cases of 99.7 M, a death toll of 2.14 M, and counting4. To date, Pakistan has received more than a million cases with a death count of over twenty-five thousand5. In a country like Pakistan, the burden on intensive care is substantial. So any intervention, before the patient lands in critical care units will greatly decrease the workload on the already saturated intensive care.

While the developed world has launched mass vaccination, the masses in developing countries are yet to be vaccinated. Despite the fact that vaccines have been launched in the developed world but their widespread availability in developing countries is still ambiguous6. The disease will continue to affect a larger population in the days to come so the search for new therapeutic agents must not cease. It is a fact that protective lung ventilation with low tidal volumes decreases mortality, off-label use of effective therapeutic agents that can decrease the progression to ARDS will be greatly beneficial7. There is growing evidence that ARDS secondary to Covid-19 is associated with disseminated intravascular and alveolar fibrin deposition8. Strategies to reduce mucous and fibrin plugs will greatly help patients. Nebulization of heparin may offer benefits over systemic administration because nebulization enhances delivery to the bronchial tree and the alveolar sacs and hence reduces the potential for systemic bleeding associated with intravenous administration. Moreover, heparin in nebulized form has greatly reduced levels of coagulation activation in the lungs both in animal studies and in patients with acute lung injury. As Heparin prevents further fibrin deposition but is ineffective in the removal of pre-existing fibrin plug, so early use of heparin during the course of the disease may help in limiting the complications of ARDS. Furthermore, it will also reduce the burden of patients in intensive care units. In this study, we will conduct a randomized controlled trial to see the effects of heparin in non-severe and severe COVID-19 patients to prevent progression to invasive mechanical ventilation or death.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 year or older.
2. Either gender
3. Currently admitted to hospital.
4. There is a PCR-positive sample for SARS-CoV-2 within the past 21 days. The sample can be a nasal or pharyngeal swab, sputum, tracheal aspirate, Broncho alveolar lavage, or another sample from the Patient
5. WHO Modified ordinal clinical scale 3-5

Exclusion Criteria:

1. Intubated and on mechanical ventilation, or requiring immediate intubation as per the treating clinician's assessment
2. Heparin allergy or heparin-induced thrombocytopenia
3. APTT >120 s, not due to anticoagulant therapy and does not correct with the administration of fresh frozen plasma
4. Platelet count <20 × 109 /L
5. Pulmonary bleeding or uncontrolled bleeding
6. Pregnant or might be pregnant
7. Acute brain injury that may result in long-term disability
8. Myopathy, spinal cord injury, or nerve injury or disease with a likely prolonged incapacity to breathe independently e.g. Guillain-Barre syndrome
9. Treatment limitations in place (Ceiling of care), i.e. not for intubation, not for ICU admission
10. Death is imminent or inevitable within 24 h
11. Clinician objection
12. Refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
Number of patients requiring Intubation | 28 days
  The primary outcome is number of patients Invasive Mechanical Ventilation (Endotracheal Intubation)or death, for patients who died before intubation

SECONDARY OUTCOMES:
Mortality | 28 Days
  Survival to day 28 and Survival to hospital discharge, censored at day 28
Oxygenation | 28 days
  Daily ratio of oxygen saturation by pulse oximetry to the fraction of inspired oxygen (SpO2/FiO2 ratio, highest and lowest levels)
Number of patients showing worsening or improvement on the modified WHO ordinal scale. | Day 7
  This is 8 points scale, starting from zero. Where 0 means uninfected and 8 means death.

CONTACTS AND LOCATIONS:
Overall Officials: Zafar Iqbal, FCPS, Study Chair — MTI, Lady Reading Hospital, Peshawar
Locations (1):
- Pulmonology Department, Lady Reading Hospital, Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Planned international meta-trial see NCT04635241
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Real-Time

REFERENCES:
- [Background] Lio KU, Rali P. Coagulopathy in COVID-19. Lung India. 2021 Mar;38(Supplement):S53-S57. doi: 10.4103/lungindia.lungindia_226_20. PMID 33686980
- [Background] van Haren FMP, Richardson A, Yoon HJ, Artigas A, Laffey JG, Dixon B, Smith R, Vilaseca AB, Barbera RA, Ismail TI, Mahrous RS, Badr M, De Nucci G, Sverdloff C, van Loon LM, Camprubi-Rimblas M, Cosgrave DW, Smoot TL, Staas S, Sann K, Sas C, Belani A, Hillman C, Shute J, Carroll M, Wilkinson T, Carroll M, Singh D, Page C. INHALEd nebulised unfractionated HEParin for the treatment of hospitalised patients with COVID-19 (INHALE-HEP): Protocol and statistical analysis plan for an investigator-initiated international metatrial of randomised studies. Br J Clin Pharmacol. 2021 Aug;87(8):3075-3091. doi: 10.1111/bcp.14714. Epub 2021 Jan 19. PMID 33377218
- [Background] Imran M, Khan S, Khan S, Uddin A, Khan MS, Ambade P. COVID-19 situation in Pakistan: A broad overview. Respirology. 2021 Sep;26(9):891-892. doi: 10.1111/resp.14093. Epub 2021 May 31. No abstract available. PMID 34056791
- [Background] Stilma W, Schultz MJ, Paulus F. Preventing mucus plugging in invasively ventilated intensive care unit patients-routine or personalized care and 'primum non nocere'. J Thorac Dis. 2018 Dec;10(12):E817-E818. doi: 10.21037/jtd.2018.11.128. No abstract available. PMID 30746263
- [Background] Chimenti L, Camprubi-Rimblas M, Guillamat-Prats R, Gomez MN, Tijero J, Blanch L, Artigas A. Nebulized Heparin Attenuates Pulmonary Coagulopathy and Inflammation through Alveolar Macrophages in a Rat Model of Acute Lung Injury. Thromb Haemost. 2017 Nov;117(11):2125-2134. doi: 10.1160/TH17-05-0347. Epub 2017 Nov 30. PMID 29202212
- [Background] Home - Johns Hopkins Coronavirus Resource Center. Johns Hopkins Coronavirus Resource Center 2021
- [Background] Villar J, Blanco J, Anon JM, Santos-Bouza A, Blanch L, Ambros A, Gandia F, Carriedo D, Mosteiro F, Basaldua S, Fernandez RL, Kacmarek RM; ALIEN Network. The ALIEN study: incidence and outcome of acute respiratory distress syndrome in the era of lung protective ventilation. Intensive Care Med. 2011 Dec;37(12):1932-41. doi: 10.1007/s00134-011-2380-4. Epub 2011 Oct 14. PMID 21997128